CLINICAL TRIAL: NCT03311165
Title: Risk Factors, Clinical Course, Treatment and Prognosis of Neonatal Acute Respiratory Distress Syndrome (ARDS): A Prospective, Observational Cohort Study
Brief Title: Epidemiological Study of Neonatal Acute Respiratory Distress Syndrome (ARDS)
Status: Completed | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: Daping Hospital of Army Medical University (Other); Jiulongpo No.1 People's Hospital (Other); Children's Hospital of Chongqing Medical University (Other); Lanzhou General Hospital of PLA (Other); First Affiliated Hospital of Chongqing Medical University (Other); Southwest Hospital, China (Other); Guiyang Maternal and Child Health Care Hospital (Other); Chengdu Women and Children's Center Hospital (Other); The Second Affiliated Hospital of the Army Medical University (Unknown); Zhujiang Hospital (Other); People's Liberation Army No.202 Hospital (Other); Bethune International Peace Hospital (Other); The 251st hosptital of PLA (Unknown); People's Hospital of Xinjiang Uygur Autonomous Region (Other); The Second Military Medical University Changhai Hospital (Unknown); The PLA Rocket Force general hospital (Unknown); the 252th Hospital of PLA (Unknown); Hunan Children's Hospital (Other Government); Wuhan general hospital of PLA (Unknown); Jinan general hospital of PLA (Unknown); The 306 Hospital of People's Liberation Army (Other); The 452nd hospital of PLA (Unknown); Xijing Hospital，FMMU (Unknown); 307 Hospital of PLA (Other); The 88th Hospital of PLA (Unknown); Tianjin Central Hospital of Gynecology Obstetrics (Other); Beijing 302 Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Nanfang Hospital, Southern Medical University (Other); Children's Hospital of Fudan University (Other); Shanxi Provincial Maternity and Children's Hospital (Other); the PLA General Hospital (Unknown); The 155th hosptital of PLA (Unknown); General Hospital of Xinjiang Military Area (Unknown); Guangzhou general hospital of PLA (Unknown); The 211st hospital of PLA (Unknown); First Affiliated Hospital of Harbin Medical University (Other); Maternal and Children's Healthcare Hospital of Taian (Other); Zhengzhou Children's Hospital, China (Other); Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); Shenyang General Hospital of PLA (Unknown); The First Affiliated Hospital of Anhui Medical University (Other); Yan'an Affiliated Hospital of Kunming Medical University (Other); Inner Mongolia People's Hospital (Other); Women and Children's Hospital, Branch of Chongqing Sanxia Central Hospital (Other); Children's Hospital of Nanjing Medical University (Other); The First Hospital of Jilin University (Other); Shanghai Children's Medical Center (Other); Ningbo Women & Children's Hospital (Other); Shandong Maternal and Child Health Hospital (Unknown); Guilin Medical College (Other); Women and Children Hospital of Qinghai Province (Other); Quanzhou Children's Hospital (Other); Newborn Department of Ankang City Central Hospital of Shaanxi Province (Unknown); the Second Hospital of Xian Jiao Tong University (Unknown); The Second Hospital of Shandong University (Other); Hunan Maternal and Children Health Hospital (Unknown); The First People's Hospital of Yinchuan (Other); The First Affiliated Hospital of Zhengzhou University (Other); The People's Hospital of Dehong Autonomous Prefecture (Other); First people Hospital of Kashi (Unknown); General Hospital of Tibet Military Region (Unknown); Navy General Hospital, Beijing (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Jiangxi Province Children's Hospital (Other); the Maternal and Child Health Hospital of Hainan Province (Other); Zhang Ye Pepole Hospital of HeXi University (Unknown); Shaanxi Provincial People's Hospital (Other); Hospital (T.C.M）Affiliated to Southwest Medical University (Unknown); Tongji Medical College,Huazhong University of Science &Techonlogy (Unknown); South Paris University Hospitals (Unknown)
Responsible Party: Principal Investigator, Ma Juan, Principal Investigator, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: 201726
Record Dates: First submitted 2017-10-04; First posted 2017-10-17 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Neonatal Acute Respiratory Distress Syndrome(ARDS)
Keywords: neonate; Acute Respiratory Distress Syndrome; prognosis; risk factor; clinical course
MeSH Terms: conditions — Respiratory Distress Syndrome; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention was given

SUMMARY:
Neonatal acute respiratory distress syndrome(ARDS) is a rare but often severe respiratory disorder. The incidence remains unclear and mortality is about 30%-60%. It is characterized by acute, refractory hypoxemia, persistent respiratory distress and decreased lung compliance. Evaluation and comparison of various clinical studies conducted were hindered by a lack of uniformity in diagnostic criteria.

DETAILED DESCRIPTION:
In 2017, the neonatal acute respiratory distress syndrome(ARDS) Consortium Working Group has proposed diagnostic criteria for neonatal ARDS. The study consists of a prospective, multicentre, web-based,cohort study in China in which neonates who fulfil the new criteria definition are enrolled in order to: describe the epidemiology, clinical course, and prognosis of neonates affected by neonatal ARDS; identify a list of risk factors for neonatal ARDS, as it exists for adults and older children with ARDS; and guide future studies.

ELIGIBILITY:
Inclusion Criteria:

* Acute onset (ie, within one week) from a known or suspected clinical insult
* Exclusion criteria: RDS, TTN, or congenital anomalies as a primary current acute respiratory condition
* Diffuse, bilateral, and irregular opacities or infiltrates, or complete opacification of the lungs, which are not fully explained by local effusions, atelectasis, RDS, TTN, or congenital anomalies
* Absence of congenital heart disease explaining the oedema (this includes ductus arteriosus with pulmonary overflow if no acute pulmonary haemorrhage exists). Echocardiography is needed to verify the origin of oedema.
* Mild ARDS: 4≤OI<8;Moderate ARDS: 8≤OI<16;Severe ARDS: OI≥16

Exclusion Criteria:

* Hyaline Membrane Disease defined as:

Mandatory criteria : defined as respiratory distress syndrome appearing within the first 24 hours of life, with response to surfactant and / or volume recruitment. Additional criteria : Lung imaging Supporting the diagnosis and / or lamellar body counts < 30,000 / mm3.

* Transient tachypnea of the neonate (wet lung) defined as:

Mandatory criteria : defined as mild ( Silverman score ≤3 ) respiratory distress appearing within the first 24 hours of life and ending within the first 48 hours of life, needing only oxygen administration and / or CPAP. Additional criteria : Lung imaging Supporting the diagnosis and / or lamellar body counts > 30,000 / mm3.

- Patients beyond the first month of life

Ages: 1 Minute to 1 Month | Sex: All
Age Groups: Child
Study Population: the definition of neonatal ARDS applies to infants from birth until 44 weeks, post-menstrual age or until 4 weeks, postnatal age (for neonates born after 40 weeks, post-menstrual age) to account for the role of prematurity; ARDS in infants older than these age limits should be diagnosed according to PALICC definition
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
bronchopulmonary dysplasia(BPD) | before discharge or 36 weeks' gestational age
  the incidence of BPD in infants with neonatal ARDS

SECONDARY OUTCOMES:
risk factors for ARDS | before discharge or 36 weeks' gestational age
  to determine risk factors leading to ARDS
death | before discharge or 36 weeks' gestational age
  the mortality in infants with neonatal ARDS
epidemiological characteristics in infants with neonatal ARDS | before discharge or 36 weeks' gestational age
  to describe the epidemiological characteristics in infants with neonatal ARDS
intraventricular hemorrhage（IVH） | before discharge or 36 weeks' gestational age
  the incidence of IVH in infants with neonatal ARDS
retinopathy of prematurity(ROP) | before discharge or 36 weeks' gestational age
  the incidence of ROP in infants with neonatal ARDS
sepsis | before discharge or 36 weeks' gestational age
  the incidence of sepsis in infants with neonatal ARDS
bronchopulmonary dysplasia(BPD) and/or death | before discharge or 36 weeks' gestational age
  the incidence of BPD and/or death in infants with neonatal ARDS
necrotizing enterocolitis(NEC) | before discharge or 36 weeks' gestational age
  the incidence of NEC in infants with neonatal ARDS

CONTACTS AND LOCATIONS:
Overall Officials: Shi Yuan, PhD,MD, Principal Investigator — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (2):
- China (2):
  - Department of Pediatrics, Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen L, Li J, Shi Y; Chinese Neonatal ARDS (ChiNARDS) study group. Clinical characteristics and outcomes in neonates with perinatal acute respiratory distress syndrome in China: A national, multicentre, cross-sectional study. EClinicalMedicine. 2022 Nov 12;55:101739. doi: 10.1016/j.eclinm.2022.101739. eCollection 2023 Jan. PMID 36386029